CLINICAL TRIAL: NCT04672200
Title: Improving Physical Activity of Older People in Community Through Trained Volunteers: the ImPACt Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Brendoncare (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 52967
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Sedentary Behavior
Keywords: Older adults; Physical activity; Group exercise; Community clubs
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): This group will receive the weekly group exercise which will be delivered online initially, and in the community clubs once they are allowed to reconvene according to government guidance. The duration of the intervention is 12 weeks.
  Interventions: Other: Group exercise

INTERVENTIONS:
Other: Group exercise — Weekly group exercises delivered online and face to face

SUMMARY:
Research question is can volunteers be trained to deliver an exercise programme for community-dwelling older people attending community clubs and is the intervention acceptable to older people and volunteers? Physical activity is important for older adults and studies have shown the benefits of physical activity on health outcomes including maintenance of physical function, improvement in well-being and quality of life, and reduction in mortality risk. A recent report on physical activity guidelines published by the Department of Health and Social Care highlighted the importance of physical activity in healthy ageing. Nonetheless, current evidence suggests that less than 7% of community-dwelling older adults meet the recommended physical activity guideline of 150 minutes of moderate vigorous physical activity per week. A review of current literature suggests some evidence that volunteers can be trained to deliver physical activity interventions for community-dwelling older people. Yet few studies have been conducted in the UK, and there is a knowledge gap in understanding the facilitators and barriers of training volunteers to deliver physical activity interventions for community-dwelling older people.

This study aims to explore the feasibility and acceptability of implementing volunteer-led exercise classes at local community clubs to encourage older people living in the community to be more active. The investigators aim to develop and evaluate a training programme for volunteers, determine the acceptability of the intervention through qualitative methods and identify facilitators and barriers to its implementation. The investigators will also explore the impact of the intervention on health outcomes for older people to inform future trial.

DETAILED DESCRIPTION:
Study design

A quasi-experimental mixed methods approach will be used to determine the feasibility and acceptability of implementing volunteer-led exercise sessions in community clubs. This feasibility study will be conducted at community-clubs managed by Brendoncare. The acceptability of the intervention will also be examined through qualitative interviews and focus groups to explore the views and experiences of volunteers and older adults involved in this study. The impact of the intervention on physical activity levels and functional outcomes will be measured.

Method

A quasi-experimental mixed methods approach will be used to determine the feasibility and acceptability of this volunteer-led physical activity intervention. This feasibility study will be conducted at community-clubs with a focus on social interactions managed by Brendoncare. Due to the Covid-19 outbreak, the community clubs are currently meeting online. The exercise intervention will be conducted online and will consist mainly of seated exercises. The impact of the intervention on physical activity levels and functional outcomes will be measured. The acceptability of the intervention will also be examined through qualitative interviews and focus groups to explore the views and experiences of volunteers and older adults involved in this study. Facilitators and barriers to the intervention will be identified to inform future implementation studies.

Participants

Community-dwelling older adults who attend Brendoncare community clubs will be invited to participate in this study. The inclusion criteria are community-dwelling older adults age 65 years and above who able to provide written consent. Club members who are not able to transfer or walk independently, and those who are actively participating in other exercise classes, will be excluded from the study. A sample size of 30 participants was chosen for pragmatic reasons for this feasibility study. Each Brendoncare club consists of between 10 - 20 regular members and to achieve the desired sample size, the intervention will need to be implemented in three clubs. The regional manager and club volunteers of the respective clubs will inform eligible club members about the study and those who are keen to participate in this study will be approached by the research team to be recruited to the study. Club members who have been approached but decline to take part will be asked if they are willing to discuss their reasons for doing so. This will help in the evaluation of the acceptability of the intervention. Due to the Covid-19 pandemic, the community clubs are currently meeting online. The clubs will reconvene according to government guidance taking into consideration social distancing measures.

Recruitment and training of volunteers

The Brendoncare clubs are managed by paid staff members but the activities are led by volunteers. Existing volunteers who are actively involved in the clubs will be invited to participate in this study and receive training to deliver the intervention. Volunteers will be provided with participant information sheets and written consent will be obtained from volunteers who are willing to participate in this study. The volunteer training programme will consist of a half a day theoretical training session followed by practical sessions. This will be conducted online. It will be led by a senior physiotherapist, Esther Clift (EC) and the study PI, Stephen Lim (SL). The training programme will be developed based on clinical expertise from therapists and current evidence including experience from a recently completed study (the SoMoVe study). The training session will include training on personal safety and safety of participants, and the exercise and mobility protocols. As these are existing volunteers, they would have been recruited, and received the generic clearance and training provided by Brendoncare. Throughout the study period, fidelity checks will be conducted by EC and SL to ensure that the volunteers are delivering high quality exercise sessions. Volunteers will also receive training on how to document adverse events that occur during the exercise classes.

Intervention

The intervention consists of a once weekly volunteer-led group exercise which will take place online and at the community clubs over 6 months. Besides exercising, participants are also encouraged to increase mobility levels. The exercise sessions will be piloted in one club before being extended to other clubs.

Data collection

Participant characteristics including age, gender, domicile status, body mass index, co-morbidities and number of medications will be recorded. PRISMA 7 will be used to characterise participants' frailty status. Mini-mental state examination (MMSE) will be used to assess participants' cognitive function. The club location, size, usual activity details and age range of club members will also be recorded to provide contextual information for each club.

The primary outcome of this study is the feasibility of implementing volunteer-led exercise sessions in the community for older adults. This will be assessed by determining the number of volunteers recruited, trained and retained at the end of the study, the number of physical activity sessions delivered and fidelity of volunteer delivery of and participants' participation in the exercise sessions. The secondary outcome measures include the measurement of physical activity levels and physical function. Physical activity levels will be measured using the CHAMPS questionnaire. Physical function will be measured using the Barthel Index. Other outcome measures include EuroQOL as a measure of quality of life, and measure of sarcopenia using SARC-F questionnaire. These outcome measures will be recorded at recruitment and repeated at 6 months and 12 months to capture any changes. Cost analysis will be conducted to determine the cost of implementing this intervention. To determine the safety of the intervention, adverse events that occur as a result of the intervention will be recorded.

Acceptability of the intervention

Interviews will be conducted among older adults and volunteers to determine the acceptability of the intervention and explore any barriers and enablers to participation and adherence to the intervention.

Older adults will be selected by purposive sampling to share their thoughts and views regarding the implementation of the volunteer-led physical activity session. To ensure a wide range of views are included in the interviews, participants will be selected to ensure equal distribution of male and female patients, different clubs and a representative age range. The aim is to interview at least three participants per club, with a total number of 9 participants.

Interviews will also be conducted for volunteers leading the intervention. The shared experience of volunteers in delivering the intervention will be explored through a group setting. The aim is to interview at least two volunteers from each club, with a total number of six volunteers.

The interviews will be semi-structured and consist of several key open-ended questions that help define the areas explored but allow the interviewer or interviewee to expand and diverge with the aim of pursuing or developing an idea with more depth. The interview schedules will be underpinned by Normalisation Process Theory.The interviews will seek to explore the views of older adults and volunteers on the exercise sessions, the barriers and facilitators to the intervention and suggestions for future implementation studies. The interviews will be audio-recorded for data collection purposes.

Data analysis

Quantitative data analysis Data collected will be double entered into a secured database for analysis. Statistical analysis will be conducted using the statistical software SPSS. Descriptive statistics -median (IQR); mean (SD); number (%) - will be used to analyse the numbers of volunteers recruited, trained and retained, as well as the type and extent of progression of the resistance exercise, and duration of their activity, and patients' adherence to the intervention. Analysis of the above outcome measures will be used to develop an assessment of the feasibility of delivering this intervention. To determine suitability for a future, fully-powered effectiveness study of the intervention, outcome measures recorded at baseline will be compared to measurement at 6 and 12 months to determine if PA intervention had an impact of physical activity levels measured by CHAMPS, functional outcomes including Barthel Index, and quality of life (EuroQol). The distribution of each outcome measure will be assessed for normality and described using parametric or non-parametric statistics accordingly. A basic cost-analysis of the training programme will be carried out, costing the time of clinical staff involved in delivering the training.

Qualitative data analysis Data collected from the interviews will be transcribed verbatim and analysed using thematic analysis (TA). The audio-recordings will be transcribed by an administrative colleague within the research department who is experienced in transcribing qualitative data. Analysis of qualitative data will be conducted using either Microsoft Word, or with the help of NVIVO, depending on the amount of data collected. Transcribed text will be read and coded separately and then together by two researchers. The codes will be analysed to generate concepts and ideas to determine the acceptability of the intervention, and to identify facilitators and barriers to the implementation process. The codes act as tags or labels to help catalogue key concepts embedded within the raw data. From the codes, themes will be developed to reflect the views and experiences of the community-dwelling older adults and volunteers regarding the community-based PA intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 year and above
* Able to walk with or without a walking aid

Exclusion Criteria:

* Attends existing exercise classes

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Volunteer training | 6 months
  The number of volunteers recruited to the study, trained and retained at the end of the study period.

SECONDARY OUTCOMES:
Physical activity levels | 6 and 12 months
  Community Healthy Activities Model Program for Seniors (CHAMPS) Physical activity questionnaire. Outcome: hours spent per week in sedentary, light, moderate and vigorous physical activity levels.
Quality of life measure | 6 and 12 months
  Measure Quality of life with EuroQol questionnaire (EQ-5D-5L), score between 0 and 100, higher score better quality life
Physical Function | 6 and 12 months
  Barthel Index, score between 0 to 100, with a higher score indicating better physical function.
Sarcopenia | 6 and 12 months
  SARC-F. Strength, Assistance with walking, Rise from a chair, Climb stairs and Falls questionnaire. The scores range from 0-10, with a higher score indicating higher risk of sarcopenia.

OTHER OUTCOMES:
Volunteer intervention | 2 months after the intervention has started.
  The acceptability of the volunteer intervention will be explored through qualitative interviews. Older adults and their careers, and volunteers will be interviewed to determine the acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lim, PhD, Principal Investigator — University of Southampton
Locations (1):
- Academic Geriatric Medicine, University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data generated from the study will be uploaded to the university repository (PURE).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years
Access Criteria: Upon request from the university.

REFERENCES:
- [Background] Lim SER, Cox NJ, Tan QY, Ibrahim K, Roberts HC. Volunteer-led physical activity interventions to improve health outcomes for community-dwelling older people: a systematic review. Aging Clin Exp Res. 2021 Apr;33(4):843-853. doi: 10.1007/s40520-020-01556-6. Epub 2020 Apr 30. PMID 32356136
- [Derived] Lim SER, Meredith SJ, Agnew S, Clift E, Ibrahim K, Roberts HC. Volunteer-led online group exercise for community-dwelling older people: a feasibility and acceptability study. BMC Geriatr. 2023 Jul 28;23(1):461. doi: 10.1186/s12877-023-04184-7. PMID 37507667
- [Derived] Lim SER, Meredith S, Agnew S, Clift E, Ibrahim K, Roberts H. Evaluating the feasibility and acceptability of virtual group exercise for older adults delivered by trained volunteers: the ImPACt study protocol. BMJ Open. 2022 Feb 1;12(2):e052631. doi: 10.1136/bmjopen-2021-052631. PMID 35105576